CLINICAL TRIAL: NCT05535530
Title: The Effect of a Newly Designed Presurgical Orthopedic Appliance on Maxillary Arch Dimensions in Infants With Bilateral Cleft Lip and Palate: Randomized Clinical Trial
Brief Title: The Effect of a Newly Designed Presurgical Orthopedic Appliance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Mushriq F. Abid, Professor, University of Baghdad
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 262421
Record Dates: First submitted 2022-08-04; First posted 2022-09-10 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Cleft Lip and Palate
Keywords: Cleft lip and palate; Bilateral; Presurgical orthopaedic appliance
MeSH Terms: conditions — Cleft Lip

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (No Intervention): Passive PSIO will be used
- Experimental (Experimental): Active PSIO will be used
  Interventions: Device: Active PSIO

INTERVENTIONS:
Device: Active PSIO — new designed active orthopedic appliance will be used. Impressions will be taken before starting the treatment (T1) and at the end of treatment (T2) three months later. The effectiveness of the two appliances will be assessed and measured on digital models of the maxillary arch before and after the treatment.
  Arms: Experimental

SUMMARY:
A randomized clinical trial to compare the effectiveness of newly designed active type of presurgical orthopedic appliances on maxillary arch dimensions in infants with bilateral cleft lip and palate.

DETAILED DESCRIPTION:
It is a multicenter randomized clinical trial with two parallel arms. The patients will be randomly divided into two groups, group one: a passive orthopedic appliance will be used, and group two a new designed active orthopedic appliance will be used. Impressions will be taken before starting the treatment (T1) and at the end of treatment (T2) three months later. The effectiveness of the two appliances will be assessed and measured on digital models of the maxillary arch before and after the treatment.

ELIGIBILITY:
Inclusion Criteria:

* 1. Healthy new born infants with complete bilateral cleft lip, alveolus and palate.

  2. Non-syndromic. 3. Non-operated cases.

Exclusion Criteria:

* 1. Infants with systemic syndromes. 2.Facial deformities.

Ages: 5 Days to 2 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-08-15 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Arch dimension (experimental group and control group) | T1 before starting any treatment and T2 After treatment before surgical repair (average 3 months)
  Evaluation of the efficiency of a newly designed presurgical infant orthopedic for bilateral cleft lip and palate patients by measuring the maxillary arch dimension at the beginning and end of treatment in both experimental and control group.

SECONDARY OUTCOMES:
Parents Perception and experience | T1 before starting any treatment and T2 After treatment before surgical repair (average 3 months)
  The perception and experience of parents of children with cleft lip and palate concerning the use presurgical infant orthopedics using a questionnaire-based cross sectional survey. The assessment of mothers' perception and experience regarding PSIO will be executed using 16 validated preformed questions. The onset of the sign of the positive correction of the cleft segments will be recorded accordingly. In addition, PSIO management, including the removable appliance's hygiene maintenance, was also assessed.
Linear measurement (experimental group and control group) | T1 before starting any treatment and T2 After treatment before surgical repair (average 3 months)
  The linear measurements of arch dimensions in millimeter before and after treatment with the new presurgical infant orthopedic within the cleft patients in both experimental and control group.
  Linear measurements for maxillary arch assessments in millimeters:
  * Antero-posterior arch length (I-RTLT)
  * Posterior arch width (RT-LT)
  * Alveolar cleft widths (AP); Right: RP-RA and left: LP-LA
  * Mid-palatal arch width (RM-LM)
Angular measurement (experimental group and control group) | T1 before starting any treatment and T2 After treatment before surgical repair (average 3 months)
  The angular measurements of arch dimensions before and after treatment with the new presurgical infant orthopedic within the cleft patients in both experimental and control group.
  Angular measurements for maxillary arch assessments in degrees:
  * Vertical deviation amount of premaxilla
  * Horizontal deviation amount of premaxilla
Vertical measurement (experimental group and control group) | T1 before starting any treatment and T2 After treatment before surgical repair (average 3 months)
  The vertical measurements of arch dimensions in millimeter before and after treatment with the new presurgical infant orthopedic within the cleft patients in both experimental and control group.
  Vertical measurements for maxillary arch assessments in millimeters:
  * The height of alveolar bone at RM
  * The height of alveolar bone at LM

CONTACTS AND LOCATIONS:
Locations (1):
- Mushreq Abed, Baghdad, Al-Rusafa, Iraq

IPD SHARING:
Plan to Share IPD: No